CLINICAL TRIAL: NCT06281054
Title: Risk and Clinical Outcomes of Acute Myocardial Infarction in Patients With Cancer: A Nationwide Study
Brief Title: Acute Myocardial Infarction in Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Associate Professor, Samsung Medical Center
Other Study IDs: SMC2023-12-027
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acute Myocardial Infarction; Cancer
Keywords: Acute myocardial infarction; Cancer; Incidence; Prognosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Revascularized Group: Cancer patients with diagnosis of acute myocardial infarction that was treated with PCI or CABG
  Interventions: Procedure: Revascularization
- Medical Group: Cancer patients with diagnosis of acute myocardial infarction that was treated with medical treatment only

INTERVENTIONS:
Procedure: Revascularization — Performing PCI or CABG
  Groups: Revascularized Group

SUMMARY:
Using national health insurance service database, current study aim to evaluate the risk and prognosis of acute myocardial infarction in cancer patients and to find the optimal treatment strategy for acute myocardial infarction that can improve long-term prognosis.

DETAILED DESCRIPTION:
This study will be conducted using Korean National Health Insurance Service database. Patients who were diagnosed with cancer from 2002 to 2021 will be included in the study. Using the selected patients, current study will analyze the incidence and prognosis of acute myocardial infarction in cancer patients and the prognosis according to the treatment method for acute myocardial infarction will be compared. Primary outcome will be all-cause death. Secondary outcomes will be myocardial infarction, revascularization, hospitalization for heart failure, stroke, and clinically relevant bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer between 2002 and 2021
* Patients who were diagnosed with acute myocardial infarction after cancer diagnosis

Exclusion Criteria:

* Patients who died during period of cancer diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with cancer from 2002 to 2021 will be considered in the study. Among these patients, those diagnosed with acute myocardial infarction after the diagnosis with cancer will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4500000 (Estimated)
Dates: Start 2002-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 2-years after diagnosis of acute myocardial infarction
  All-cause death which was obtained from death certification collected by Statistics Korea at the Ministry of Strategy and Finance of South Korea

SECONDARY OUTCOMES:
Myocardial infarction | 2-years after diagnosis of acute myocardial infarction
  Myocardial infarction is defined as presence of the diagnostic codes (ICD-10 I21, I22) in the primary position during hospitalization
Revascularization | 2-years after diagnosis of acute myocardial infarction
  Percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
Hospitalization for heart failure | 2-years after diagnosis of acute myocardial infarction
  Heart failure events requiring hospitalization defined as presence of the diagnostic codes (I110, I130, I132, I255, I420, I425-I429, I43, I50, I971) in the primary position during hospitalization
Stroke | 2-years after diagnosis of acute myocardial infarction
  Stroke is defined as ischemic stroke (ICD-10 I63, I64) or intracranial hemorrhage (ICD-10 I60-62), combined with the codes of diagnostic brain imaging.
Clinically relevant bleeding | 2-years after diagnosis of acute myocardial infarction
  Bleeding requiring hospitalization or transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center; Seung Hun Lee, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Chonnam National University Medical School, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No
This is National Health Insurance Data Analysis. Therefore, sharing the original patient-level data is not possible under regulation by the Korean government.